CLINICAL TRIAL: NCT04725188
Title: A Phase 2, Multicenter, Randomized Study to Compare the Efficacy and Safety of MK-7684A or MK-7684A Plus Docetaxel Versus Docetaxel Monotherapy in the Treatment of Participants With Metastatic Non-small Cell Lung Cancer With Progressive Disease After Treatment With a Platinum Doublet Chemotherapy and Immunotherapy
Brief Title: Pembrolizumab/Vibostolimab Coformulation (MK-7684A) or Pembrolizumab/Vibostolimab Coformulation Plus Docetaxel Versus Docetaxel for Metastatic Non Small Cell Lung Cancer (NSCLC) With Progressive Disease After Platinum Doublet Chemotherapy and Immunotherapy (MK-7684A-002, KEYVIBE-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7684A-002; MK-7684A-002 (Other: MSD); KEYVIBE-002 (Other: MSD); 2022-501252-28-00 (Registry Identifier: EU CT); U1111-1275-8661 (Registry Identifier: UTN); 2020-004034-38 (EudraCT Number)
Record Dates: First submitted 2021-01-25; First posted 2021-01-26 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Non Small Cell Lung Cancer
Keywords: Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); Programmed Cell Death Receptor Ligand 2 (PD-L2); PD-1; PDL1; PD-L1; PD-L2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Arm 1 and Arm 3: Double-blind with in-house blinding Arm 2: Unblinded Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Pembrolizumab/Vibostolimab coformulation + Docetaxel (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous (IV) infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years plus docetaxel 75 mg/m^2 via IV infusion Q3W. Each cycle will be 21 days.
  Interventions: Biological: Pembrolizumab/Vibostolimab coformulation; Drug: Docetaxel
- Arm 2: Pembrolizumab/Vibostolimab coformulation (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via IV infusion Q3W for up to 35 cycles up to approximately 2 years. Each cycle will be 21 days.
  Interventions: Biological: Pembrolizumab/Vibostolimab coformulation
- Arm 3: Placebo + Docetaxel (Active Comparator): Participants receive normal saline placebo via IV infusion Q3W for up to 35 cycles up to approximately 2 years plus docetaxel 75 mg/m^2 IV infusion Q3W. Each cycle will be 21 days.
  Interventions: Drug: Docetaxel; Drug: Placebo

INTERVENTIONS:
Biological: Pembrolizumab/Vibostolimab coformulation — Pembrolizumab 200 mg + vibostolimab 200 mg/20 mL vial IV infusion Q3W up to approximately 2 years.
  Other Names: MK-7684A
  Arms: Arm 1: Pembrolizumab/Vibostolimab coformulation + Docetaxel; Arm 2: Pembrolizumab/Vibostolimab coformulation
Drug: Docetaxel — Docetaxel 75 mg^m2 IV infusion Q3W until discontinuation due to progressive disease or unacceptable toxicity. Docetaxel will serve as part of an experimental treatment in Arm 1, and as an active comparator in Arm 3.
  Other Names: Taxotere
  Arms: Arm 1: Pembrolizumab/Vibostolimab coformulation + Docetaxel; Arm 3: Placebo + Docetaxel
Drug: Placebo — Normal saline IV infusion Q3W up to approximately 2 years
  Arms: Arm 3: Placebo + Docetaxel

SUMMARY:
The main purpose of this study is to compare pembrolizumab/vibostolimab coformulation (MK-7684A) plus docetaxel or pembrolizumab/vibostolimab coformulation to normal saline placebo plus docetaxel. Participants with metastatic non-small cell lung cancer (NSCLC) and progressive disease (PD) after platinum doublet chemotherapy and treatment with one prior anti- programmed cell death 1 (PD-1)/ programmed cell death ligand 1(PD-L1) monoclonal antibody (mAb). MK-7684A is a coformulation product of pembrolizumab/vibostolimab. The dual primary hypotheses of the study are pembrolizumab/vibostolimab coformulation plus docetaxel and pembrolizumab/vibostolimab coformulation is superior to normal saline placebo plus docetaxel with respect to progression free survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by blinded independent central review (BICR).

DETAILED DESCRIPTION:
Participants may receive additional 17 cycles of pembrolizumab/vibostolimab (each cycle length = 21 days) for an additional 1 year of treatment as second course phase at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of metastatic non-small cell lung cancer (NSCLC)
* Has confirmation that epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), or reactive oxygen species (ROS) 1 directed therapy is not indicated as primary therapy
* Has progressive disease (PD) on treatment with one prior anti-programmed cell death 1 (PD-1)/ programmed cell death ligand 1 (PD-L1) monoclonal antibody (mAb) administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies

  * Retreatment with the same anti-PD-L1/PD-L1 mAb is acceptable in the overall course of treatment
* Has PD as determined by the investigator after platinum doublet chemotherapy for metastatic disease
* Has measurable disease defined as at least 1 measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI), based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
* Has provided tumor tissue for PD-L1 biomarker analysis from an archival sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Has a life expectancy of at least 3 months
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1 assessed within 7 days prior to randomization
* Male participants randomized to docetaxel are eligible to participant if they agree to refrain from donating sperm, and either 1) be abstinent from heterosexual intercourse; or 2) must agree to follow contraceptive guidance as per study protocol unless confirmed to be azoospermic during the intervention period and for at least 180 days after the last dose of docetaxel
* Female participants must be not pregnant, not breastfeeding, and not be a woman of child-bearing potential (WOCBP). A WOCBP is eligible is she agrees to either use contraception, or be abstinent from heterosexual intercourse during the intervention period and for ≥120 days after the last dose of study intervention. If a WOCBP is randomized to docetaxel, she agrees not to donate eggs and either uses contraception or be abstinent from heterosexual intercourse during the treatment period and for ≥180 days after the last dose of docetaxel
* Has adequate organ function

Exclusion Criteria:

* Has known active or untreated central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for at least 3 years since initiation of that therapy
* Has received docetaxel as monotherapy or in combination with other therapies
* Has received previous treatment with another agent targeting the T-cell immunoreceptor with immunoglobulin [Ig] and immunoreceptor tyrosine-based inhibitory motif [ITIM] domains (TIGIT) pathway
* Has received radiotherapy within 2 weeks of start of study intervention. One week washout is permitted for palliative radiation to non-CNS disease
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention
* Has severe hypersensitivity (≥Grade 3) to docetaxel or pembrolizumab/vibostolimab coformulation and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of study intervention
* Has interstitial lung disease, or history of pneumonitis requiring steroids for treatment
* Has known history of active human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C
* Has had an allogenic tissue/solid organ transplant
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (95):
- United States (10):
  - Cedars-Sinai Medical Center ( Site 2522), Los Angeles, California
  - Illinois Cancer Care ( Site 2534), Peoria, Illinois
  - Baptist Health Lexington-Research ( Site 2502), Lexington, Kentucky
  - University of Maryland ( Site 2528), Baltimore, Maryland
  - Hattiesburg Clinic Hematology/Oncology ( Site 2511), Hattiesburg, Mississippi
  - Mercy Research - Cancer and Hematology Center ( Site 2535), Springfield, Missouri
  - Mercy Research - David C. Pratt Cancer Center ( Site 2532), St Louis, Missouri
  - Montefiore- Einstein Center for Cancer Care-Oncology ( Site 2509), The Bronx, New York
  - University of Cincinnati Medical Center-University of Cincinnati Cancer Center ( Site 2526), Cincinnati, Ohio
  - St Francis Cancer Center-Research Office ( Site 2531), Greenville, South Carolina
- Argentina (6):
  - Centro de Oncología e Investigación de Buenos Aires ( Site 0008), Berazategui, Buenos Aires
  - Hospital Privado de Comunidad ( Site 0004), Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0002), Mar del Plata, Buenos Aires
  - Instituto de Oncología de Rosario ( Site 0003), Rosario, Santa Fe Province
  - Hospital Privado Universitario de Córdoba ( Site 0001), Córdoba
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 0005), La Rioja
- Australia (3):
  - Canberra Hospital ( Site 0104), Canberra, Australian Capital Territory
  - Gold Coast University Hospital-Clinical Trials Service ( Site 0106), Southport, Queensland
  - Fiona Stanley Hospital-Medical Oncology ( Site 0102), Murdoch, Western Australia
- Austria (3):
  - Medizinische Universität Graz ( Site 0201), Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen-Department of Pneumology ( Site 0203), Linz, Upper Austria
  - Klinik Floridsdorf-Abteilung für Innere Medizin und Pneumologie ( Site 0204), Vienna
- Belgium (5):
  - AZ Sint-Maarten, Campus Leopoldstraat 2 ( Site 0333), Mechelen, Antwerpen
  - UZ Brussel ( Site 0336), Brussels, Bruxelles-Capitale, Region de
  - Grand Hôpital de Charleroi-Oncology & Hematology ( Site 0337), Charleroi, Hainaut
  - Jessa Ziekenhuis-Pulmonology & Thoracic Oncology ( Site 0338), Hasselt, Limburg
  - AZ Nikolaas ( Site 0334), Sint-Niklaas, Oost-Vlaanderen
- Brazil (4):
  - Hospital Nossa Senhora da Conceição ( Site 0403), Porto Alegre, Rio Grande do Sul
  - ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO-Pesquisa Clinica ( Site 0400), São Paulo, São Paulo
  - Centro de Tratamento de Tumores Botafogo - CTTB-Pesquisa Clínica ( Site 0402), Rio de Janeiro
  - Hospital Paulistano ( Site 0406), São Paulo
- Denmark (3):
  - Rigshospitalet ( Site 0702), Copenhagen, Capital Region
  - Odense Universitetshospital ( Site 0700), Odense, Region Syddanmark
  - Sygehus Soenderjylland-Kraeftambulatoriet ( Site 0705), Sønderborg, Region Syddanmark
- Finland (4):
  - Oulun yliopistollinen sairaala ( Site 0902), Oulu, North Ostrobothnia
  - Tampereen yliopistollinen sairaala-Oncology ( Site 0906), Tampere, Pirkanmaa
  - Vaasan Keskussairaala ( Site 0903), Vaasa, Pohjanmaa
  - Turku University Hospital-The Department of Pulmonary Medicine ( Site 0905), Turku, Southwest Finland
- France (9):
  - Nouvel Hôpital Civil (NHC) ( Site 1000), Strasbourg, Alsace
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cance-Medical Oncology ( Site 1009), Bordeaux, Aquitaine
  - Centre Hospitalier Universitaire de Caen - Hôpital Côte de Nacre ( Site 1006), Caen, Calvados
  - CHU de Toulouse - Hopital Larrey-service de pneumologie ( Site 1008), Toulouse, Haute-Garonne
  - Clinique Ambroise Paré ( Site 1007), Beuvry, Pas-de-Calais
  - Centre Hospitalier du Mans ( Site 1002), Le Mans, Sarthe
  - Gustave Roussy ( Site 1005), Villejuif, Val-de-Marne
  - HIA Sainte Anne ( Site 1003), Toulon, Var
  - Centre Hospitalier d'Avignon-Service d'Oncologie médicale et d'hématologie clinique ( Site 1004), Avignon, Vaucluse
- Germany (5):
  - Onkologie Ravensburg ( Site 1104), Ravensburg, Baden-Wurttemberg
  - Klinikverbund Allgaeu gGmbH ( Site 1109), Immenstadt im Allgäu, Bavaria
  - Helios Dr. Horst Schmidt Kliniken ( Site 1108), Wiesbaden, Hesse
  - Universitätsklinikum Bonn ( Site 1111), Bonn, North Rhine-Westphalia
  - Helios Klinikum Emil von Behring Berlin-Zehlendorf ( Site 1106), Berlin
- Israel (4):
  - Soroka Medical Center ( Site 1202), Beersheba
  - Rambam Health Care Campus-Oncology ( Site 1203), Haifa
  - Shaare Zedek Medical Center-Oncology ( Site 1206), Jerusalem
  - Sourasky Medical Center ( Site 1205), Tel Aviv
- Italy (8):
  - Azienda Ospedaliera S. Giovanni Addolorata-Oncologia Medica ( Site 1307), Rome, Lazio
  - Azienda Ospedaliera Dei Colli-U.O.C Pneumologia Oncologica DH PNL ONC ( Site 1308), Naples, Napoli
  - CRO-IRCCS-medical oncology ( Site 1304), Aviano, Pordenone
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga-Oncologia Polmonare ( Site 1300), Orbassano, Torino
  - Azienda Ospedaliera Universitaria Careggi-SOD ONCOLOGIA MEDICA ( Site 1306), Florence, Tuscany
  - Ospedale San Raffaele-Oncologia Medica ( Site 1305), Milan
  - Istituto Europeo di Oncologia IRCCS-Divisione di Oncologia Toracica ( Site 1301), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli-Medical Oncology ( Site 1303), Roma
- Malaysia (4):
  - Hospital Sultan Ismail ( Site 1503), Johor Bahru, Johor
  - University Malaya Medical Centre ( Site 1501), Lembah Pantai, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan ( Site 1500), Kuantan, Pahang
  - Beacon Hospital Sdn Bhd ( Site 1504), Petaling Jaya, Selangor
- Poland (2):
  - Przychodnia Lekarska KOMED ( Site 1704), Konin, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier, Warsaw, Masovian Voivodeship
- Russia (9):
  - Saint Petersburg State University-Clinic of advanced medical technologies n. a. Nicolay I. Pirogov (, Saint Petersburg, Leningradskaya Oblast'
  - Saint-Petersburg City Clinical Oncology Dispensary-Department of chemotherapy ( Site 1911), Saint Petersburg, Leningradskaya Oblast'
  - Moscow Clinical Research Center-Chemotherapy department ( Site 1910), Moscow, Moscow
  - Central Clinical Hospital of the Presidential Administrative Department ( Site 1902), Moscow, Moscow
  - Hadassah Medical-Oncology department ( Site 1912), Moscow, Moscow Oblast
  - Nizhegorodsky Regional Oncology Dispensary, Branch #2-chemotherapy ( Site 1909), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Budgetary Healthcare Institution of Omsk Region Clinical Oncology Dispensary ( Site 1908), Omsk, Omsk Oblast
  - GBUZ LOKB-Oncology department #1 ( Site 1905), Saint Petersburg, Sankt-Peterburg
  - N.N.Petrov Research Institute of Oncology-Department of Chemotherapy and Innovative Technologies ( S, Saint Petersburg, Sankt-Peterburg
- South Korea (4):
  - Seoul National University Bundang Hospital ( Site 2003), Seongnam, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital-Medical Oncology ( Site 2005), Suwon, Kyonggi-do
  - Chungbuk National University Hospital-Internal medicine ( Site 2004), Cheongju-si, North Chungcheong
  - Asan Medical Center-Oncology ( Site 2000), Songpagu, Seoul
- Spain (4):
  - HOSPITAL CLÍNIC DE BARCELONA-ICHMO- Clinic Institut of Haematological and Oncological diseases ( Sit, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau-Oncología Médica ( Site 2102), Barcelona, Catalonia
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON-ONCOLOGY ( Site 2101), Madrid
  - Hospital Universitario Virgen de Valme-Departamento de Oncologia ( Site 2103), Seville
- Ospedale Regionale Bellinzona e Valli ( Site 2203), Bellinzona, Canton Ticino, Switzerland
- Taiwan (5):
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 2303), Kaohsiung Niao Sung Dist, Kaohsiung
  - Taichung Veterans General Hospital-Chest ( Site 2307), Taichung
  - NATIONAL CHENG-KUNG UNI. HOSP.-clinical trial center ( Site 2302), Tainan
  - National Taiwan University Hospital-Oncology ( Site 2304), Taipei
  - Mackay Memorial Hospital-Chest Medicine ( Site 2305), Taipei
- Thailand (2):
  - Chulalongkorn University ( Site 2403), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 2400), Bangkok, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26206&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel: Participants received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous (IV) infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years plus docetaxel 75 mg/m^2 via IV infusion Q3W. Each cycle was 21 days.
- Arm 2: Pembrolizumab/Vibostolimab Coformulation: Participants received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via IV infusion Q3W for up to 35 cycles up to approximately 2 years. Each cycle was 21 days.
- Arm 3: Placebo + Docetaxel: Participants received normal saline placebo via IV infusion Q3W for up to 35 cycles up to approximately 2 years plus docetaxel 75 mg/m^2 via IV infusion Q3W. Each cycle was 21 days.
Period: Overall Study
Arm/Group | Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel | Arm 2: Pembrolizumab/Vibostolimab Coformulation | Arm 3: Placebo + Docetaxel
Started | 87 | 83 | 85
Treated | 85 | 83 | 83
Completed | 0 | 0 | 0
Not Completed | 87 | 83 | 85
Not completed — Death | 72 | 69 | 76
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Sponsor Decision | 12 | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel | Arm 2: Pembrolizumab/Vibostolimab Coformulation | Arm 3: Placebo + Docetaxel | Total
Number analyzed (Participants) | 87 | 83 | 85 | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (8.8) | 66.0 (7.4) | 65.8 (8.0) | 65.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 24 | 74
  Male | 60 | 60 | 61 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 6 | 27
  Not Hispanic or Latino | 62 | 68 | 65 | 195
  Unknown or Not Reported | 13 | 6 | 14 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 14 | 10 | 35
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 1 | 2
  White | 62 | 63 | 60 | 185
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 13 | 5 | 14 | 32
Programmed Cell Death Ligand 1 (PD-L1) Status at Baseline [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a biopsy. Randomization of participants in the study was stratified by PD-L1 tumor proportion score (TPS) at baseline (<1%, 1-49%, or ≥ 50%). Higher percentages of PD-L1 TPS staining correspond to higher positivity of PD-L1 on a tumor. Participants were classified as follows: <1% = PD-L1 negative, 1-49% = PD-L1 weakly positive; and ≥50% = PD-L1 strongly positive.
  Participants
    Tumor proportion score (TPS) ≥50% | 15 | 14 | 13 | 42
    TPS 1-49% | 34 | 19 | 35 | 88
    TPS <1% | 37 | 45 | 34 | 116
    Unknown (Not evaluable due to <100 viable tumor cells) | 1 | 5 | 3 | 9
Predominant Tumor Histology [Count of Participants; unit: Participants] — Participants were classified according to tumor histology: Squamous or Non-squamous.
  Participants
    Squamous | 26 | 20 | 34 | 80
    Non-squamous | 61 | 63 | 51 | 175
Prior Lines of Therapy [Count of Participants; unit: Participants] — Participants were classified according to the number of prior lines of therapy they received to treat their metastatic Non Small Cell Lung Cancer (NSCLC): 1, 2, 3, 4, or ≥5.
  Participants
    1 | 58 | 49 | 52 | 159
    2 | 25 | 28 | 26 | 79
    3 | 1 | 4 | 7 | 12
    4 | 1 | 2 | 0 | 3
    ≥5 | 2 | 0 | 0 | 2
Sequence of Prior Anti-Programmed Cell Death Receptor 1 (PD-1)/PD-L1 [Count of Participants; unit: Participants] — Participants were stratified by the timing of prior Anti-PD-1/PD-L1 therapy: immediate prior therapy versus not immediate prior therapy.
  Participants
    Immediate Prior Therapy | 72 | 70 | 72 | 214
    Not the Immediate Prior Therapy | 15 | 13 | 13 | 41
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  Participants
    ECOG = 0 | 34 | 30 | 32 | 96
    ECOG = 1 | 53 | 53 | 53 | 159

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) Assessment
Description: PFS is defined as the time from randomization to the first documented disease progression (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR is presented.
Time Frame: Up to approximately 21 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel | Arm 2: Pembrolizumab/Vibostolimab Coformulation | Arm 3: Placebo + Docetaxel
Number analyzed (Participants) | 87 | 83 | 85
Months | 5.6 [3.9 to 6.8] | 2.7 [1.8 to 4.0] | 3.2 [2.8 to 5.7]
Statistical Analysis 1: Comparison: Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel vs Arm 3: Placebo + Docetaxel; Test type: Superiority; p = 0.0910, Regression, Cox; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.53 to 1.13]
Statistical Analysis 2: Comparison: Arm 2: Pembrolizumab/Vibostolimab Coformulation vs Arm 3: Placebo + Docetaxel; Test type: Superiority; p = 0.9622, Regression, Cox; Hazard Ratio (HR) = 1.40, 95% CI 2-sided [0.96 to 2.02]

2. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 by BICR Assessment
Description: ORR is defined as the percentage of participants who have a confirmed complete response (CR: Disappearance of all target lesions) or a partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR as assessed by BICR based on RECIST 1.1 is presented.
Time Frame: Up to approximately 21 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel | Arm 2: Pembrolizumab/Vibostolimab Coformulation | Arm 3: Placebo + Docetaxel
Number analyzed (Participants) | 87 | 83 | 85
Percentage of participants | 29.9 [20.5 to 40.6] | 6.0 [2.0 to 13.5] | 15.3 [8.4 to 24.7]
Statistical Analysis 1: Comparison: Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel vs Arm 3: Placebo + Docetaxel; Test type: Superiority; p = 0.0113, Miettinen & Nurminen method; Difference in percentage = 14.7, 95% CI 2-sided [2.1 to 26.9]
Statistical Analysis 2: Comparison: Arm 2: Pembrolizumab/Vibostolimab Coformulation vs Arm 3: Placebo + Docetaxel; Test type: Superiority; p = 0.9750, Miettinen & Nurminen method; Difference in percentage = -9.4, 95% CI 2-sided [-19.6 to 0.0]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to the date of death due to any cause.
Time Frame: Up to approximately 21 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel | Arm 2: Pembrolizumab/Vibostolimab Coformulation | Arm 3: Placebo + Docetaxel
Number analyzed (Participants) | 87 | 83 | 85
Months | 10.2 [8.6 to 14.9] | 7.5 [5.2 to 13.4] | 8.8 [6.4 to 11.1]
Statistical Analysis 1: Comparison: Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel vs Arm 3: Placebo + Docetaxel; Test type: Superiority; p = 0.0943, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.50 to 1.15]
Statistical Analysis 2: Comparison: Arm 2: Pembrolizumab/Vibostolimab Coformulation vs Arm 3: Placebo + Docetaxel; Test type: Superiority; p = 0.5974, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.70 to 1.58]

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 by BICR Assessment
Description: For participants who demonstrate a confirmed CR (Disappearance of all target lesions) or confirmed PR (At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until disease progression (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. The DOR as assessed by BICR is presented.
Time Frame: Up to approximately 21 months
Population: All randomized participants who demonstrated a confirmed CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel | Arm 2: Pembrolizumab/Vibostolimab Coformulation | Arm 3: Placebo + Docetaxel
Number analyzed (Participants) | 26 | 5 | 13
Months | 6.5 [5.3 to 10.7] | NA [2.8 to NA] — NA=Median DOR not reached at time of data cutoff due to insufficient number of responding participants with relapse NA=DOR upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse | NA [3.0 to NA] — NA = Median DOR not reached at time of data cutoff due to insufficient number of responding participants with relapse NA=DOR upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced an AE is reported here.
Time Frame: Up to approximately 39 months
Population: Per protocol, the safety analysis population consisted of all randomized participants who received at least 1 dose of study treatment. Participants are included in the treatment group corresponding to the study treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel | Arm 2: Pembrolizumab/Vibostolimab Coformulation | Arm 3: Placebo + Docetaxel
Number analyzed (Participants) | 85 | 83 | 83
Participants | 85 | 76 | 82

6. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment due to an AE is reported here.
Time Frame: Up to approximately 27 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Pembrolizumab/Vibostolimab Coformulation + Docetaxel | Arm 2: Pembrolizumab/Vibostolimab Coformulation | Arm 3: Placebo + Docetaxel
Number analyzed (Participants) | 85 | 83 | 83
Participants | 42 | 12 | 24

ADVERSE EVENTS:
Time Frame: Up to approximately 39 months
Description: All-cause mortality included all randomized participants. Serious and other AEs included all randomized participants who received at least 1 dose of study treatment. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Groups:
- Pembrolizumab/Vibostolimab Coformulation + Docetaxel: Participants received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous (IV) infusion once every 3 weeks (Q3W) for up to 35 cycles up to approximately 2 years plus docetaxel 75 mg/m^2 via IV infusion Q3W. Each cycle was 21 days.
- Pembrolizumab/Vibostolimab Coformulation: Participants received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via IV infusion Q3W for up to 35 cycles up to approximately 2 years. Each cycle was 21 days.
- Placebo + Docetaxel: Participants received normal saline placebo via IV infusion Q3W for up to 35 cycles up to approximately 2 years plus docetaxel 75 mg/m^2 via IV infusion Q3W. Each cycle was 21 days.
Arm/Group | Pembrolizumab/Vibostolimab Coformulation + Docetaxel | Pembrolizumab/Vibostolimab Coformulation | Placebo + Docetaxel
All-Cause Mortality (participants affected / at risk) | 74/87 | 70/83 | 77/85
Serious Adverse Events (participants affected / at risk) | 48/85 | 26/83 | 37/83
Other Adverse Events (participants affected / at risk) | 83/85 | 67/83 | 76/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab/Vibostolimab Coformulation + Docetaxel (N=85) | Pembrolizumab/Vibostolimab Coformulation (N=83) | Placebo + Docetaxel (N=83)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (3)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Segmental diverticular colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 7 (9) | 3 (3) | 10 (11)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subperiosteal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Lichenification (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Euthanasia (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab/Vibostolimab Coformulation + Docetaxel (N=85) | Pembrolizumab/Vibostolimab Coformulation (N=83) | Placebo + Docetaxel (N=83)
Anaemia (Blood and lymphatic system disorders) | 30 (35) | 12 (13) | 28 (30)
Hyperthyroidism (Endocrine disorders) | 5 (6) | 2 (2) | 2 (2)
Hypothyroidism (Endocrine disorders) | 8 (10) | 3 (3) | 1 (1)
Lacrimation increased (Eye disorders) | 7 (7) | 0 (0) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 2 (2) | 6 (6)
Constipation (Gastrointestinal disorders) | 20 (28) | 6 (6) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 31 (52) | 10 (12) | 23 (33)
Nausea (Gastrointestinal disorders) | 24 (38) | 11 (12) | 22 (26)
Stomatitis (Gastrointestinal disorders) | 14 (23) | 1 (1) | 5 (7)
Vomiting (Gastrointestinal disorders) | 12 (16) | 4 (5) | 11 (16)
Asthenia (General disorders) | 26 (38) | 15 (16) | 24 (28)
Chest pain (General disorders) | 2 (2) | 4 (4) | 6 (6)
Fatigue (General disorders) | 26 (39) | 10 (10) | 23 (26)
Mucosal inflammation (General disorders) | 6 (10) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 17 (21) | 3 (3) | 8 (9)
Pyrexia (General disorders) | 7 (7) | 5 (7) | 11 (15)
COVID-19 (Infections and infestations) | 13 (14) | 6 (6) | 7 (7)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6) | 6 (7)
Amylase increased (Investigations) | 3 (3) | 5 (8) | 1 (2)
Blood creatinine increased (Investigations) | 5 (5) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 2 (3) | 5 (8) | 1 (1)
Neutrophil count decreased (Investigations) | 14 (25) | 0 (0) | 15 (24)
Weight decreased (Investigations) | 14 (16) | 4 (4) | 11 (12)
Decreased appetite (Metabolism and nutrition disorders) | 21 (28) | 11 (11) | 19 (25)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (9) | 2 (2) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 3 (3) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (6) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (22) | 3 (3) | 11 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (14) | 1 (1) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (9) | 2 (2) | 5 (7)
Dysgeusia (Nervous system disorders) | 12 (13) | 0 (0) | 7 (9)
Headache (Nervous system disorders) | 5 (5) | 3 (4) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 14 (15) | 0 (0) | 7 (7)
Paraesthesia (Nervous system disorders) | 4 (5) | 1 (1) | 6 (7)
Insomnia (Psychiatric disorders) | 8 (8) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 5 (5) | 11 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 14 (15) | 14 (14)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (24) | 2 (2) | 20 (21)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (9) | 2 (2) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 4 (4)
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (5)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 31 (51) | 17 (21) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 22 (28) | 15 (17) | 7 (8)
Hypertension (Vascular disorders) | 5 (6) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT04725188/Prot_SAP_001.pdf